CLINICAL TRIAL: NCT04002245
Title: A Pilot Study, Non-comparative Efficiency of Techniques of 'Snail ' and 'Go-back' Application of an Alcoholic Antiseptic on Healthy Skin Before the Placement of a Intra-vascular Device,
Brief Title: A Pilot Study Efficiency of Techniques of 'Snail ' and 'Go-back' Application of an Alcoholic Antiseptic on Healthy Skin Before the Placement of a Intra-vascular Device,
Acronym: TApAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2018/36
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Health Care Utilization
Keywords: vascular access; skin antisepsis; cutaneous antisepsis
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: From the paper randomisation list that has been communicated to him, he learns the application technique to be performed on each of the two arms (right or left).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Go back (Experimental): Application of a compress impregnated with alcoholic Betadine® by movement of return
  Interventions: Procedure: antiseptic application
- Technique of snail (Experimental): Application of a compress impregnated with alcoholic Betadine into a single movement from the center towards the periphery and covering the end surface of followed by spontaneous drying time 30 seconds.
  Interventions: Procedure: antiseptic application

INTERVENTIONS:
Procedure: antiseptic application — The application of the antiseptic on the healthy and visibly clean skin of the bend of the elbow will be carried out for all participant

SUMMARY:
Given the lack of scientific data on the effect of the antiseptic application technique on reducing the number of microorganisms present during application, this pilot study will provide data on the initial level of microorganisms in this population of healthy volunteers and on the difference before and after antiseptic application according to both techniques. These data will be useful to then calculate the study size suitable for a formal comparative study.

DETAILED DESCRIPTION:
During their care, many patients benefit from invasive procedures. These treatments involve a break-in of the healthy skin which, without the application of preventive measures, can be at the origin of an infection starting from the micro-organisms present on the skin.

Cutaneous antisepsis, which objective is to reduce or even eliminate commensal and transient flora microorganisms, is an essential preventive measure during an invasive act on healthy skin. The choice of antiseptic most suitable in this context has been the subject of numerous publications and recommendations (including: French Society of Hospital Hygiene - SF2H- 2016). But there is no consensus on application technique.

In France, there is two application techniques : the "snail" and the "back and forth" techniques. These two techniques have never been compared in clinical trials. This study will bring preliminary evidence on empirical practices, in order to complement the recommendations of good antiseptic practices and ultimately reduce infections.

This brings us to the following question: what are the effects of the application of an alcoholic antiseptic by "back and forth" and "snail" techniques on healthy skin? We'll conduced a monocentric non-comparative, randomized, matched pilot study, to provide data on the initial level of microorganisms in this population of healthy volunteers and on the difference before and after antiseptic application according to both techniques. These data will be useful to then calculate the study size suitable for a formal comparative study between application techniques.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Nursing student (NS)
* Signed consent
* Major (18 years old and over)

Exclusion Criteria:

* Allergy to the antiseptic used in the study
* Contamination visible at the bend of the elbow
* Impossibility to carry out the procedure on one of the arms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Number of microorganisms | Day 1
  Average difference in the number of microorganisms between the initial and final samples.

CONTACTS AND LOCATIONS:
Overall Officials: Yolène CARRE, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- ISFI Pellegrin - CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No